CLINICAL TRIAL: NCT04063215
Title: A Clinical Trial to Determine the Safety and Efficacy of Hope Biosciences Autologous Mesenchymal Stem Cell Therapy for the Treatment of Traumatic Brain Injury and Hypoxic-Ischemic Encephalopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hope Biosciences LLC (Industry)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Organization: Hope Biosciences Research Foundation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBTBI01
Record Dates: First submitted 2019-08-13; First posted 2019-08-21 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury
Keywords: severe; hypoxic-ischemic encephalopathy; stroke; intracranial hemorrhage; cerebral palsy; chronic; neurological injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Lymphoma, Follicular; Hypoxia-Ischemia, Brain; Stroke; Intracranial Hemorrhages; Cerebral Palsy; Bronchiolitis Obliterans Syndrome; Trauma, Nervous System

STUDY DESIGN:
Intervention Model Description: Single arm, non-randomized study to determine safety and treatment effect of three infusions of HB-adMSC (2 x 10^8 total cells per dose) in adult patients with sub-acute or chronic neurological injury
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HB-adMSC (Experimental): HB-adMSCs will be infused three times spaced 14 days apart (Week 0, Week 2, Week 4)
  Interventions: Biological: HB-adMSCs

INTERVENTIONS:
Biological: HB-adMSCs — Hope Biosciences autologous adipose-derived mesenchymal stem cells

SUMMARY:
This study aims to determine the safety of HB-adMSC infusion and treatment effects of HB-adMSC infusion on brain structure, neurocognitive/functional outcomes, and neuroinflammation after subacute and chronic neurological injury in adults.

DETAILED DESCRIPTION:
This study aims to determine the safety of HB-adMSC infusion and treatment effects of HB-adMSC infusion on global gray and/or white matter, as well as structural integrity of GM and WM regions of interest in the corpus callous and corticospinal tracts as measured by fractional anisotropy (FA) and mean diffusivity (MD) in specific regions known to correlate with specific neurocognitive deficits in patients after neurological injury.

ELIGIBILITY:
Inclusion Criteria:

1. adults between 18 and 55 years of age
2. documented head injury with functional neurological damage to the central nervous system unlikely to improve with present standard of care approaches
3. a Glasgow Outcome Scale-Extended (GOS-E) score > 2 and ≤ 6
4. onset or diagnosis of the injury or disease process greater than 6 months
5. ability to obtain consent from the subject of their legally authorized representative (LAR)
6. ability to speak English or Spanish *required for validated neurocognitive outcome testing) -

Exclusion Criteria:

1. known history of:

   1. intellectual deficiency or psychiatric conditions likely to invalidate our ability to assess changes in cognition or behavior,
   2. recently treated infection,
   3. renal disease or altered renal function (screening serum creatinine > 1.5 mg/dL),
   4. hepatic disease or altered liver function (screening SGPT > 150 U/L or T. Bilirubin >1.3 mg/dL),
   5. cancer,
   6. immunosuppression (screening WBC < 3, 000 cells/ml),
   7. HIV+,
   8. chemical or ETOH dependency that in the opinion of the investigator would preclude participation in the study,
   9. acute or chronic lung disease requiring significant medication, oxygen supplementation, or mechanical ventilation,
   10. bleeding disorders including immune-mediated heparin-induced thrombocytopenia,
   11. known sensitivity to heparin, Lovenox, and pork products,
   12. individuals with mechanical prosthetic heart valves.
   13. individuals who have received a stem cell treatment.
2. Normal brain CT/MRI exam
3. Spinal deformity, spinal surgery (including repeated epidural or spinal punctures), or spinal cord injury diagnosed by CT/MR or clinical exam
4. diagnosed with a genetic or metabolic disorder related to the neurologic condition
5. other acute or chronic medical conditions that, in the opinion of the investigator, may increase the risks associated with study participation
6. for women of child bearing potential, a positive pregnancy test at the screening visit, or, for both women and men, unwillingness to comply with acceptable methods of birth control during the study
7. participation in a concurrent interventional study
8. inability to undergo the diagnostic tests (PET/DT-MRI) or unwilling/unable to cooperate with the diagnostic tests and outcome assessments
9. unwilling or unable to return for follow-up study visits -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles S Cox, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital-Clinical Research Unit (MMH-CRU), Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: HB-adMSCs will be infused three times over a six week period, spaced 14 days apart
  HB-adMSCs: Hope Biosciences autologous adipose-derived mesenchymal stem cells
Period: Overall Study
Arm/Group | Treatment Group
Started | 24
Completed | 20
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: Autologous Hope Biosciences adipose derived mesenchymal stem cells. HB-adMSCs: HB-adMSCs will be administered intravenously to study participants who qualify.
  Placebo: Placebo will be administered intravenously to study participants who qualify.
Arm/Group | Treatment Group
Number analyzed (Participants) | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 73 (19)
Height [Mean (Standard Deviation); unit: cm] | 175 (14)
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (10)
Age, Customized [Median (Inter-Quartile Range); unit: Years] | 33 [27 to 41]

OUTCOME MEASURES:

1. Primary Outcome: Vital Signs (Respiratory Rate)
Description: Mean and Standard Deviation of Vital Signs at Visits 1, 3, 6, and 7 for Respiratory Rate
Time Frame: Screening/Pre-Infusion (Visit 1), Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56)
Population: Some subjects either withdrew or were lost to follow-up before specific time points of the study, causing slight variation of subject population between visits. Additionally, some subjects missed various assessments at different points of the study.
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
breaths/min
  Screening/Pre-Infusion (Visit 1) | 16.54 (1.22)
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 22
  Infusion 1/Baseline (Visit 3 - Week 0) | 16.82 (1.59)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 20
  6 months Post-Infusion (Visit 6 - Week 28) | 16.63 (0.96)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 19
  1 year Post-Infusion (Visit 7 - Week 56) | 16.42 (0.84)

2. Primary Outcome: Vital Signs (Temperature)
Description: Mean and Standard Deviation of Vital Signs at Visits 1, 3, 6, and 7 for Temperature
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
degrees Celsius
  Screening/Pre-Infusion (Visit 1) | 36.76 (0.55)
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 22
  Infusion 1/Baseline (Visit 3 - Week 0) | 42.49 (18.18)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 20
  6 months Post-Infusion (Visit 6 - Week 28) | 39.85 (13.68)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 19
  1 year Post-Infusion (Visit 7 - Week 56) | 39.96 (14.08)

3. Primary Outcome: Vital Signs (Systolic Blood Pressure)
Description: Mean and Standard Deviation of Vital Signs at Visits 1, 3, 6, and 7 for Systolic Blood Pressure
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
mmHg
  Screening/Pre-Infusion (Visit 1) | 119 (16)
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 22
  Infusion 1/Baseline (Visit 3 - Week 0) | 119 (14)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 20
  6 months Post-Infusion (Visit 6 - Week 28) | 117 (14)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 19
  1 year Post-Infusion (Visit 7 - Week 56) | 119 (14)

4. Primary Outcome: Vital Signs (Diastolic Blood Pressure)
Description: Mean and Standard Deviation of Vital Signs at Visits 1, 3, 6, and 7 for Diastolic Blood Pressure
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
mmHg
  Screening/Pre-Infusion (Visit 1) | 73 (9)
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 22
  Infusion 1/Baseline (Visit 3 - Week 0) | 72 (8)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 20
  6 months Post-Infusion (Visit 6 - Week 28) | 74 (10)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 19
  1 year Post-Infusion (Visit 7 - Week 56) | 74 (8)

5. Primary Outcome: Vital Signs (Pulse Rate)
Description: Mean and Standard Deviation of Vital Signs at Visits 1, 3, 6, and 7 for Pulse Rate
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
beats/min
  Screening/Pre-Infusion (Visit 1) | 80 (12)
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 22
  Infusion 1/Baseline (Visit 3 - Week 0) | 78 (9)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 20
  6 months Post-Infusion (Visit 6 - Week 28) | 80 (16)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 19
  1 year Post-Infusion (Visit 7 - Week 56) | 76 (13)

6. Primary Outcome: Vital Signs (Oxygen Saturation)
Description: Mean and Standard Deviation of Vital Signs at Visits 1, 3, 6, and 7 for Oxygen Saturation
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of oxygen
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
% of oxygen
  Screening/Pre-Infusion (Visit 1) | 98.87 (1.60)
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 22
  Infusion 1/Baseline (Visit 3 - Week 0) | 98.68 (1.84)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 20
  6 months Post-Infusion (Visit 6 - Week 28) | 98.37 (1.74)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 19
  1 year Post-Infusion (Visit 7 - Week 56) | 98.79 (1.25)

7. Primary Outcome: Vital Signs Change From Baseline (Diastolic Blood Pressure)
Description: Mean and Standard Deviation of Vital Signs Change from Baseline at Visits 3, 4, and 5 for Diastolic Blood Pressure
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0), Infusion 2 (Visit 4 - Week 2), Infusion 3 (Visit 5 - Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
mmHg
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 22
  Infusion 1/Baseline (Visit 3 - Week 0) | 71.0 (10.42)
  Infusion 2 (Visit 4 - Week 2): number analyzed (Participants) | 22
  Infusion 2 (Visit 4 - Week 2) | 69.4 (10.24)
  Infusion 2 (Visit 4 - Week 2) Change from Baseline: number analyzed (Participants) | 22
  Infusion 2 (Visit 4 - Week 2) Change from Baseline | -1.7 (8.69)
  Infusion 3 (Visit 5 - Week 4): number analyzed (Participants) | 22
  Infusion 3 (Visit 5 - Week 4) | 68.8 (9.31)
  Infusion 3 (Visit 5 - Week 4) Change from Baseline: number analyzed (Participants) | 22
  Infusion 3 (Visit 5 - Week 4) Change from Baseline | -2.1 (8.81)

8. Primary Outcome: Vital Signs Change From Baseline (Systolic Blood Pressure)
Description: Mean and Standard Deviation of Vital Signs Change from Baseline at Visits 3, 4, and 5 for Systolic Blood Pressure
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0), Infusion 2 (Visit 4 - Week 2), Infusion 3 (Visit 5 - Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
mmHg
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 22
  Infusion 1/Baseline (Visit 3 - Week 0) | 115.3 (14.73)
  Infusion 2 (Visit 4 - Week 2): number analyzed (Participants) | 22
  Infusion 2 (Visit 4 - Week 2) | 113.8 (16.06)
  Infusion 2 (Visit 4 - Week 2) Change from Baseline: number analyzed (Participants) | 22
  Infusion 2 (Visit 4 - Week 2) Change from Baseline | -1.7 (11.10)
  Infusion 3 (Visit 5 - Week 4): number analyzed (Participants) | 22
  Infusion 3 (Visit 5 - Week 4) | 114.3 (15.18)
  Infusion 3 (Visit 5 - Week 4) Change from Baseline: number analyzed (Participants) | 22
  Infusion 3 (Visit 5 - Week 4) Change from Baseline | -1.0 (11.18)

9. Primary Outcome: Vital Signs Change From Baseline (Pulse Rate)
Description: Mean and Standard Deviation of Vital Signs Change from Baseline at Visits 3, 4, and 5 for Pulse Rate
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0), Infusion 2 (Visit 4 - Week 2), Infusion 3 (Visit 5 - Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
beats/min
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 22
  Infusion 1/Baseline (Visit 3 - Week 0) | 72.0 (11.26)
  Infusion 2 (Visit 4 - Week 2): number analyzed (Participants) | 22
  Infusion 2 (Visit 4 - Week 2) | 70.5 (11.15)
  Infusion 2 (Visit 4 - Week 2) Change from Baseline: number analyzed (Participants) | 22
  Infusion 2 (Visit 4 - Week 2) Change from Baseline | -1.4 (10.79)
  Infusion 3 (Visit 5 - Week 4): number analyzed (Participants) | 22
  Infusion 3 (Visit 5 - Week 4) | 72.1 (11.02)
  Infusion 3 (Visit 5 - Week 4) Change from Baseline: number analyzed (Participants) | 22
  Infusion 3 (Visit 5 - Week 4) Change from Baseline | 0.1 (11.15)

10. Primary Outcome: Vital Signs Change From Baseline (Oxygen Saturation)
Description: Mean and Standard Deviation of Vital Signs Change from Baseline at Visits 3, 4, and 5 for Oxygen Saturation
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0), Infusion 2 (Visit 4 - Week 2), Infusion 3 (Visit 5 - Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of oxygen
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
% of oxygen
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 22
  Infusion 1/Baseline (Visit 3 - Week 0) | 97.1 (4.63)
  Infusion 2 (Visit 4 - Week 2): number analyzed (Participants) | 22
  Infusion 2 (Visit 4 - Week 2) | 97.5 (1.97)
  Infusion 2 (Visit 4 - Week 2) Change from Baseline: number analyzed (Participants) | 22
  Infusion 2 (Visit 4 - Week 2) Change from Baseline | 0.4 (4.59)
  Infusion 3 (Visit 5 - Week 4): number analyzed (Participants) | 22
  Infusion 3 (Visit 5 - Week 4) | 96.7 (5.15)
  Infusion 3 (Visit 5 - Week 4) Change from Baseline: number analyzed (Participants) | 22
  Infusion 3 (Visit 5 - Week 4) Change from Baseline | -0.5 (6.82)

11. Primary Outcome: Vital Signs Change From Baseline (Respiratory Rate)
Description: Mean and Standard Deviation of Vital Signs Change from Baseline at Visits 3, 4, and 5 for Respiratory Rate
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0), Infusion 2 (Visit 4 - Week 2), Infusion 3 (Visit 5 - Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
breaths/min
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 22
  Infusion 1/Baseline (Visit 3 - Week 0) | 16.4 (1.67)
  Infusion 2 (Visit 4 - Week 2): number analyzed (Participants) | 22
  Infusion 2 (Visit 4 - Week 2) | 16.4 (1.14)
  Infusion 2 (Visit 4 - Week 2) Change from Baseline: number analyzed (Participants) | 22
  Infusion 2 (Visit 4 - Week 2) Change from Baseline | 0.0 (1.40)
  Infusion 3 (Visit 5 - Week 4): number analyzed (Participants) | 22
  Infusion 3 (Visit 5 - Week 4) | 16.4 (1.03)
  Infusion 3 (Visit 5 - Week 4) Change from Baseline: number analyzed (Participants) | 22
  Infusion 3 (Visit 5 - Week 4) Change from Baseline | 0.0 (1.83)

12. Primary Outcome: Vital Signs Change From Baseline (Temperature)
Description: Mean and Standard Deviation of Vital Signs Change from Baseline at Visits 3, 4, and 5 for Temperature
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0), Infusion 2 (Visit 4 - Week 2), Infusion 3 (Visit 5 - Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
degrees Celsius
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 22
  Infusion 1/Baseline (Visit 3 - Week 0) | 36.7 (0.29)
  Infusion 2 (Visit 4 - Week 2): number analyzed (Participants) | 22
  Infusion 2 (Visit 4 - Week 2) | 36.7 (0.25)
  Infusion 2 (Visit 4 - Week 2) Change from Baseline: number analyzed (Participants) | 22
  Infusion 2 (Visit 4 - Week 2) Change from Baseline | 0.0 (0.35)
  Infusion 3 (Visit 5 - Week 4): number analyzed (Participants) | 22
  Infusion 3 (Visit 5 - Week 4) | 36.7 (0.29)
  Infusion 3 (Visit 5 - Week 4) Change from Baseline: number analyzed (Participants) | 22
  Infusion 3 (Visit 5 - Week 4) Change from Baseline | -0.0 (0.36)

13. Secondary Outcome: Interleukin 4
Description: IL-4 lab measure of patients from a bead-based, ELISA/Flow Cytometry combination assay to evaluate cytokine measures at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56)
  Values ranged from 1940 pg/mL to 6060 pg/mL
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
pg/mL
  Infusion 1/Baseline (Visit 3 - Week 0) | 2694 (939)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 4236 (2561)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 18
  1 year Post-Infusion (Visit 7 - Week 56) | 3388 (1296)
Statistical Analysis 1: Comparison: HB-adMSC; For inflammatory cytokines, time course data will be analyzed using a GLMM to test differences across time between pre- and post- treatment. The dependent variables will be the neuroinflammatory biomarkers with time (to model the trajectory) and GOSE (3-4 or 5-8) as covariates and a random subject effect (to account for within subject correlation). Point estimates of pre- and posttreatment differences will be reported along with 95% confidence interval; Test type: Other; p = 0.048, Mixed Models Analysis

14. Secondary Outcome: Interleukin 2
Description: IL-2 lab measure of patients from a bead-based, ELISA/Flow Cytometry combination assay to evaluate cytokine measures at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56)
  Values ranged from 363 pg/mL to 1909 pg/mL
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
pg/mL
  Infusion 1/Baseline (Visit 3 - Week 0) | 652 (221)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 828 (517)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 18
  1 year Post-Infusion (Visit 7 - Week 56) | 973 (324)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.2, Mixed Models Analysis

15. Secondary Outcome: Interleukin 1-beta
Description: IL-1-beta lab measure of patients from a bead-based, ELISA/Flow Cytometry combination assay to evaluate cytokine measures at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56)
  Values range from 1615 pg/mL to 6930 pg/mL
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
pg/mL
  Infusion 1/Baseline (Visit 3 - Week 0) | 3267 (780)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 3709 (1763)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 18
  1 year Post-Infusion (Visit 7 - Week 56) | 3478 (1226)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.6, Mixed Models Analysis

16. Secondary Outcome: Interferon Gamma-induced Protein 10 (IP-10)
Description: IP-10 lab measure of patients from a bead-based, ELISA/Flow Cytometry combination assay to evaluate cytokine measures at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56)
  Values ranged from 5270 pg/mL to 15466 pg/mL
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
pg/mL
  Infusion 1/Baseline (Visit 3 - Week 0) | 8090 (2762)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 8158 (2210)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 18
  1 year Post-Infusion (Visit 7 - Week 56) | 7426 (1828)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.10, Mixed Models Analysis

17. Secondary Outcome: Tumor Necrosis Factor Alpha
Description: TNFα lab measure of patients from a bead-based, ELISA/Flow Cytometry combination assay to evaluate cytokine measures at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56)
  Values ranged from 232 pg/mL to 4570 pg/mL
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
pg/mL
  Infusion 1/Baseline (Visit 3 - Week 0) | 1246 (775)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 1694 (1497)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 18
  1 year Post-Infusion (Visit 7 - Week 56) | 1553 (609)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.4, Mixed Models Analysis

18. Secondary Outcome: Monocyte Chemoattractant Protein-1 (MCP-1)
Description: MCP-1 lab measure of patients from a bead-based, ELISA/Flow Cytometry combination assay to evaluate cytokine measures at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56)
  Values range from 1439 pg/mL to 7472 pg/mL
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
pg/mL
  Infusion 1/Baseline (Visit 3 - Week 0) | 4600 (1602)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 4745 (1122)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 18
  1 year Post-Infusion (Visit 7 - Week 56) | 5090 (833)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.6, Mixed Models Analysis

19. Secondary Outcome: Interleukin Protein-17A (IL-17a)
Description: IL-17a lab measure of patients from a bead-based, ELISA/Flow Cytometry combination assay to evaluate cytokine measures at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56)
  Values measure 526 pg/mL to 3228 pg/mL
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
pg/mL
  Infusion 1/Baseline (Visit 3 - Week 0) | 1529 (532)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 1410 (827)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 18
  1 year Post-Infusion (Visit 7 - Week 56) | 1736 (639)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.5, Mixed Models Analysis

20. Secondary Outcome: Interleukin 6
Description: IL-6 lab measure of patients from a bead-based, ELISA/Flow Cytometry combination assay to evaluate cytokine measures at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56)
  Values range from 750 pg/mL to 4740 pg/mL
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
pg/mL
  Infusion 1/Baseline (Visit 3 - Week 0) | 1501 (574)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 1609 (1379)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 18
  1 year Post-Infusion (Visit 7 - Week 56) | 1695 (681)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 13, analysis 1]; Test type: Other; p > 0.9, Mixed Models Analysis

21. Secondary Outcome: Interleukin 10
Description: IL-10 lab measure of patients from a bead-based, ELISA/Flow Cytometry combination assay to evaluate cytokine measures at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56)
  Values range from 497 pg/mL to 2796 pg/mL
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
pg/mL
  Infusion 1/Baseline (Visit 3 - Week 0) | 1020 (388)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 1129 (777)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 18
  1 year Post-Infusion (Visit 7 - Week 56) | 1087 (337)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.8, Mixed Models Analysis

22. Secondary Outcome: IFN-gamma
Description: IFN-gamma lab measure of patients from a bead-based, ELISA/Flow Cytometry combination assay to evaluate cytokine measures at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56)
  Values range from 764 pg/mL to 6591 pg/mL
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
pg/mL
  Infusion 1/Baseline (Visit 3 - Week 0) | 1419 (826)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 2940 (1779)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 18
  1 year Post-Infusion (Visit 7 - Week 56) | 1696 (679)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.002, Mixed Models Analysis

23. Secondary Outcome: IL-12p70
Description: IL-12p70 lab measure of patients from a bead-based, ELISA/Flow Cytometry combination assay to evaluate cytokine measures at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56)
  Values range from 676 pg/mL to 3975 pg/mL
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
pg/mL
  Infusion 1/Baseline (Visit 3 - Week 0) | 1835 (385)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 1708 (1097)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 18
  1 year Post-Infusion (Visit 7 - Week 56) | 1893 (652)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.8, Mixed Models Analysis

24. Secondary Outcome: IL-8
Description: IL-8 lab measure of patients from a bead-based, ELISA/Flow Cytometry combination assay to evaluate cytokine measures at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56)
  Values range from 1348 pg/mL to 7738 pg/mL
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
pg/mL
  Infusion 1/Baseline (Visit 3 - Week 0) | 2477 (927)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 3667 (2161)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 18
  1 year Post-Infusion (Visit 7 - Week 56) | 3023 (1181)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.069, Mixed Models Analysis

25. Secondary Outcome: Free Active TGF-Beta1
Description: Free active TGF-Beta1 lab measure of patients from a bead-based, ELISA/Flow Cytometry combination assay to evaluate cytokine measures at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56)
  Values range from 799 pg/mL to 7374 pg/mL
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
pg/mL
  Infusion 1/Baseline (Visit 3 - Week 0) | 1684 (1580)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 2252 (2251)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 18
  1 year Post-Infusion (Visit 7 - Week 56) | 1755 (1244)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.6, Mixed Models Analysis

26. Secondary Outcome: Glasgow Outcome Scale-Expanded (GOS-E) Functional Outcomes
Description: Count of Participants with specific GOS-E scores at Visits 3, 6, and 7 Glasgow Outcome Scale-Extended is an 8-point scale that classifies the global outcome for individuals with traumatic brain injury (TBI), ranging from 1 (dead) to 8 (upper good recovery). The categorical rating is based on a structured interview about the patient's ability to function. Higher scores indicate better recovery. Category 3 is Lower Severe Disability, Category 4 is Upper Severe Disability, Category 5 is Lower Moderate Disability, and Category 6 is Upper Moderate Disability.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
Participants
  Category 3 at Infusion 1/Baseline (Visit 3 - Week 0) | 7
  Category 4 at Infusion 1/Baseline (Visit 3 - Week 0) | 5
  Category 5 at Infusion 1/Baseline (Visit 3 - Week 0) | 2
  Category 6 at Infusion 1/Baseline (Visit 3 - Week 0) | 10
  Category 3 at 6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 20
  Category 3 at 6 months Post-Infusion (Visit 6 - Week 28) | 6
  Category 4 at 6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 20
  Category 4 at 6 months Post-Infusion (Visit 6 - Week 28) | 3
  Category 5 at 6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 20
  Category 5 at 6 months Post-Infusion (Visit 6 - Week 28) | 2
  Category 6 at 6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 20
  Category 6 at 6 months Post-Infusion (Visit 6 - Week 28) | 9
  Category 3 at 1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 20
  Category 3 at 1 year Post-Infusion (Visit 7 - Week 56) | 5
  Category 4 at 1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 20
  Category 4 at 1 year Post-Infusion (Visit 7 - Week 56) | 2
  Category 5 at 1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 20
  Category 5 at 1 year Post-Infusion (Visit 7 - Week 56) | 3
  Category 6 at 1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 20
  Category 6 at 1 year Post-Infusion (Visit 7 - Week 56) | 10
Statistical Analysis 1: Comparison: HB-adMSC; A proportional odds logistic regression model was used to analyze the data over time. This model is used to predict an ordered categorical outcome over time by assuming the odds ratio between any two outcome categories is constant throughout all time points. Null hypothesis is that time has no effect on the cumulative odds for a patient to be in a higher category after being evaluated on the GOS-E. Odds ratio >1 indicates higher likelihood of being in higher categories compared to at baseline; Test type: Other; p = 0.63, Regression, Logistic — This p-value applies to data regarding 6 months Post-Infusion (Visit 6 - Week 28) compared to Infusion 1/Baseline (Visit 3 - Week 0); Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.43 to 4.19]; This statistical analysis applies to data regarding 6 months Post-Infusion (Visit 6 - Week 28) compared to Infusion 1/Baseline (Visit 3 - Week 0)
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 26, analysis 1]; Test type: Other; p = 0.36, Regression, Logistic — This p-value applies to data regarding 1 year Post-Infusion (Visit 7 - Week 56) compared to Infusion 1/Baseline (Visit 3 - Week 0); Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.55 to 5.45]; This statistical analysis applies to data regarding 1 year Post-Infusion (Visit 7 - Week 56) compared to Infusion 1/Baseline (Visit 3 - Week 0)

27. Secondary Outcome: Disability Rating Scale (DRS) Functional Outcomes
Description: Mean and SD of Disability Rating Scale (DRS) evaluation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The Disability Rating Scale score provides a numerical measure of an individual's functional impairment and disability. This assessment uses a 0-30 total score to assess traumatic brain injury, with higher scores indicating greater disability. A score of 0 indicates a rating of "no disability" and a score of 30 indicates a rating of "profound vegetative state".
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
score on a scale
  Infusion 1/Baseline (Visit 3 - Week 0) | 4.54 (3.89)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 20
  6 months Post-Infusion (Visit 6 - Week 28) | 4.65 (4.07)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 20
  1 year Post-Infusion (Visit 7 - Week 56) | 3.30 (2.00)
Statistical Analysis 1: Comparison: HB-adMSC; Neuropsychological and Functional outcome measures were analyzed using general linear mixed models (GLMMs) to estimate differences across time points (pre- and post-treatment). Models will include time of assessment (baseline and 6 and/or 12 months after treatment) and baseline age as covariates with random intercepts for participants to account for within-participant correlation. Mean differences with 95% confidence intervals were determined for all outcomes at 6 and 12 months after treatment; Test type: Other; p = 0.047, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.19; Mean Difference (Net) = -0.38, 95% CI 2-sided [-0.75 to -0.01] — Effect size: 0.19
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.00023, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.19; Mean Difference (Net) = -0.749, 95% CI 2-sided [-1.12 to -0.379] — Effect size: 0.19

28. Secondary Outcome: Galveston Orientation and Amnesia Test Neuropsychological Outcomes
Description: Mean and SD of Galveston Orientation and Amnesia Test (GOAT) evaluation of cognition at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The total score is calculated by subtracting an "error score" from 100. The error score is calculated by summing together the individual error score points from each question. The minimum total score of -3 is associated with a failure to respond correctly to any memory/orientation question. A total score of 100 indicates perfect recall on the GOAT memory/orientation questions. Higher total scores indicate better recall.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
score on a scale
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 23
  Infusion 1/Baseline (Visit 3 - Week 0) | 91.74 (7.81)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 95.89 (4.93)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 20
  1 year Post-Infusion (Visit 7 - Week 56) | 96.10 (4.56)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.00027, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.63; Mean Difference (Net) = 4.86, 95% CI 2-sided [2.42 to 7.29] — Effect size: 0.63
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.00019, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.63; Mean Difference (Net) = 4.9, 95% CI 2-sided [2.506 to 7.294] — Effect size: 0.63

29. Secondary Outcome: Brief Symptoms Inventory 18 (BSI 18) SOM T Scores
Description: Brief Symptoms Inventory 18 (BSI 18) Somatization (SOM) T-Score Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The BSI-18 has three subscores (somatization, depression, and anxiety) each with a raw score of 0 to 24, with higher scores indicating greater distress. A T-score is then calculated by comparing to normative data. T-scores under 50 indicate no elevation and T-scores of 63 or higher suggests a clinically significant level of distress. T-scores are standardized to have an average of 50 and a standard deviation of 10. Technically there is no minimum or maximum t-score since it is normalized.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 23
  Infusion 1/Baseline (Visit 3 - Week 0) | 56.52 (9.85)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 52.42 (8.93)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 20
  1 year Post-Infusion (Visit 7 - Week 56) | 51.60 (7.86)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.19, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.38; Mean Difference (Net) = -2.43, 95% CI 2-sided [-6.07 to -1.18] — Effect size: 0.38
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.043, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.38; Mean Difference (Net) = -3.7, 95% CI 2-sided [-7.26 to -0.14] — Effect size: 0.38

30. Secondary Outcome: Brief Symptoms Inventory 18 (BSI 18) DEP T Scores
Description: Brief Symptoms Inventory 18 (BSI 18) Depression (DEP) T-Score Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The BSI-18 has three subscores (somatization, depression, and anxiety) each with a raw score of 0 to 24, with higher scores indicating greater distress. A T-score is then calculated by comparing to normative data. T-scores under 50 indicate no elevation and T-scores of 63 or higher suggests a clinically significant level of distress. T-scores are standardized to have an average of 50 and a standard deviation of 10. Technically there is no minimum or maximum t-score since it is normalized.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 23
  Infusion 1/Baseline (Visit 3 - Week 0) | 57.17 (12.83)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 52.58 (11.65)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 20
  1 year Post-Infusion (Visit 7 - Week 56) | 51.00 (11.68)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.069, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.48; Mean Difference (Net) = -3.63, 95% CI 2-sided [-7.55 to 0.26] — Effect size: 0.48
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.026, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.48; Mean Difference (Net) = -6.15, 95% CI 2-sided [-9.983 to -2.317] — Effect size: 0.48

31. Secondary Outcome: Brief Symptoms Inventory 18 (BSI 18) Anxiety (ANX) T Scores
Description: Brief Symptoms Inventory 18 (BSI 18) Anxiety (ANX) T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The BSI-18 has three subscores (somatization, depression, and anxiety) each with a raw score of 0 to 24, with higher scores indicating greater distress. A T-score is then calculated by comparing to normative data. T-scores under 50 indicate no elevation and T-scores of 63 or higher suggests a clinically significant level of distress. T-scores are standardized to have an average of 50 and a standard deviation of 10. Technically there is no minimum or maximum t-score since it is normalized.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 23
  Infusion 1/Baseline (Visit 3 - Week 0) | 54.74 (10.85)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 48.37 (9.06)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 20
  1 year Post-Infusion (Visit 7 - Week 56) | 47.85 (8.71)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.020, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.53; Mean Difference (Net) = -4.43, 95% CI 2-sided [-8.12 to -0.79] — Effect size: 0.53
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.0029, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.53; Mean Difference (Net) = -5.7, 95% CI 2-sided [-9.297 to -2.103] — Effect size: 0.53

32. Secondary Outcome: Brief Symptoms Inventory 18 (BSI 18) Global Severity Index (GSI) T Scores
Description: Brief Symptoms Inventory 18 (BSI 18) Global Severity Index (GSI) T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The BSI-18 has three subscores (somatization, depression, and anxiety) each with a raw score of 0 to 24, with higher scores indicating greater distress. The Global Severity Index (GSI) is the sum of the three subscores, which was then normalized with a t-score in this analysis. A T-score was calculated by comparing to normative data. T-scores under 50 indicate no elevation and T-scores of 63 or higher suggests a clinically significant level of distress. T-scores are standardized to have an average of 50 and a standard deviation of 10. Technically there is no minimum or maximum t-score since it is normalized.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 23
  Infusion 1/Baseline (Visit 3 - Week 0) | 57.48 (11.14)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 52.00 (10.37)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 20
  1 year Post-Infusion (Visit 7 - Week 56) | 50.60 (10.69)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.054, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.53; Mean Difference (Net) = -3.64, 95% CI 2-sided [-7.33 to 0.02] — Effect size: 0.53
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.0023, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.53; Mean Difference (Net) = -5.85, 95% CI 2-sided [-9.456 to -2.244] — Effect size: 0.53

33. Secondary Outcome: TBI Quality of Life Questionnaires (TBI-QOL SF) - Cognition - General Concerns T Scores
Description: TBI Quality of Life Questionnaires (TBI-QOL SF) - Cognition - General Concerns T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The TBI-QOL SF consists of multiple subsections that are summed individually to create a raw score for each subsection. Then, a T-score was calculated by comparing to normative data. T-scores are standardized to have an average of 50 and a standard deviation of 10. A higher T-score indicates more of the measured construct was observed, whether it is a positive construct or a negative construct. Technically there is no minimum or maximum t-score since it is normalized. A score of 60 is above average and a score of 40 is below average.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 23
  Infusion 1/Baseline (Visit 3 - Week 0) | 37.29 (8.85)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 41.85 (7.01)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 20
  1 year Post-Infusion (Visit 7 - Week 56) | 42.72 (9.01)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.0097, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.51; Mean Difference (Net) = 3, 95% CI 2-sided [0.79 to 5.22] — Effect size: 0.51
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.00017, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.51; Mean Difference (Net) = 4.51, 95% CI 2-sided [2.335 to 6.685] — Effect size: 0.51

34. Secondary Outcome: TBI Quality of Life Questionnaires (TBI-QOL SF) - Communication T Scores
Description: TBI Quality of Life Questionnaires (TBI-QOL SF) - Communication T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The TBI-QOL SF consists of multiple subsections that are summed individually to create a raw score for each subsection. Then, a T-score was calculated by comparing to normative data. T-scores are standardized to have an average of 50 and a standard deviation of 10. A higher T-score indicates more of the measured construct was observed, whether it is a positive construct or a negative construct. Technically there is no minimum or maximum t-score since it is normalized. A score of 60 is above average and a score of 40 is below average.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 23
  Infusion 1/Baseline (Visit 3 - Week 0) | 47.76 (8.91)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 52.18 (7.08)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 20
  1 year Post-Infusion (Visit 7 - Week 56) | 52.39 (10.60)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.049, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.40; Mean Difference (Net) = 2.58, 95% CI 2-sided [0.04 to 5.14] — Effect size: 0.40
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.0069, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.40; Mean Difference (Net) = 3.555, 95% CI 2-sided [1.054 to 6.056] — Effect size: 0.40

35. Secondary Outcome: TBI Quality of Life Questionnaires (TBI-QOL SF) - Independence T Scores
Description: TBI Quality of Life Questionnaires (TBI-QOL SF) - Independence T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The TBI-QOL SF consists of multiple subsections that are summed individually to create a raw score for each subsection. Then, a T-score was calculated by comparing to normative data. T-scores are standardized to have an average of 50 and a standard deviation of 10. A higher T-score indicates more of the measured construct was observed, whether it is a positive construct or a negative construct. Technically there is no minimum or maximum t-score since it is normalized. A score of 60 is above average and a score of 40 is below average.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 23
  Infusion 1/Baseline (Visit 3 - Week 0) | 40.10 (8.82)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 43.51 (8.82)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 20
  1 year Post-Infusion (Visit 7 - Week 56) | 44.95 (7.70)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.0064, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.57; Mean Difference (Net) = 4.03, 95% CI 2-sided [1.21 to 6.82] — Effect size: 0.57
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.00076, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.57; Mean Difference (Net) = 5.005, 95% CI 2-sided [2.251 to 7.759] — Effect size: 0.57

36. Secondary Outcome: TBI Quality of Life Questionnaires (TBI-QOL SF) - Mobility T Scores
Description: TBI Quality of Life Questionnaires (TBI-QOL SF) - Mobility T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The TBI-QOL SF consists of multiple subsections that are summed individually to create a raw score for each subsection. Then, a T-score was calculated by comparing to normative data. T-scores are standardized to have an average of 50 and a standard deviation of 10. A higher T-score indicates more of the measured construct was observed, whether it is a positive construct or a negative construct. Technically there is no minimum or maximum t-score since it is normalized. A score of 60 is above average and a score of 40 is below average.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 23
  Infusion 1/Baseline (Visit 3 - Week 0) | 39.36 (11.85)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 40.12 (11.73)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 20
  1 year Post-Infusion (Visit 7 - Week 56) | 40.73 (11.30)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.0084, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.23; Mean Difference (Net) = 3.13, 95% CI 2-sided [0.86 to 5.38] — Effect size: 0.23
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.018, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.23; Mean Difference (Net) = 2.72, 95% CI 2-sided [0.5 to 4.94] — Effect size: 0.23

37. Secondary Outcome: TBI Quality of Life Questionnaires (TBI-QOL SF) - Satisfaction With SRA T Scores
Description: TBI Quality of Life Questionnaires (TBI-QOL SF) - Satisfaction with SRA T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The TBI-QOL SF consists of multiple subsections that are summed individually to create a raw score for each subsection. Then, a T-score was calculated by comparing to normative data. T-scores are standardized to have an average of 50 and a standard deviation of 10. A higher T-score indicates more of the measured construct was observed, whether it is a positive construct or a negative construct. Technically there is no minimum or maximum t-score since it is normalized. A score of 60 is above average and a score of 40 is below average.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Groups:
- HB-adMSC: HB-adMSCs will be infused three times spaced 14 days apart (Week 0, Week 2, Week 4)
  HB-adMSCs: Hope Biosciences autologous adipose-derived mesenchymal stem cell
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 23
  Infusion 1/Baseline (Visit 3 - Week 0) | 41.96 (6.50)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 44.53 (4.26)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 20
  1 year Post-Infusion (Visit 7 - Week 56) | 44.35 (5.04)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.024, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.36; Mean Difference (Net) = 2.22, 95% CI 2-sided [0.33 to 4.13] — Effect size: 0.36
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.017, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.36; Mean Difference (Net) = 2.31, 95% CI 2-sided [0.445 to 4.175] — Effect size: 0.36

38. Secondary Outcome: TBI Quality of Life Questionnaires (TBI-QOL SF) - Upper Extremity/ADL T Scores
Description: TBI Quality of Life Questionnaires (TBI-QOL SF) - Upper Extremity/ADL T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The TBI-QOL SF consists of multiple subsections that are summed individually to create a raw score for each subsection. Then, a T-score was calculated by comparing to normative data. T-scores are standardized to have an average of 50 and a standard deviation of 10. A higher T-score indicates more of the measured construct was observed, whether it is a positive construct or a negative construct. Technically there is no minimum or maximum t-score since it is normalized. A score of 60 is above average and a score of 40 is below average.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 23
  Infusion 1/Baseline (Visit 3 - Week 0) | 37.20 (10.98)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 36.65 (9.76)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 20
  1 year Post-Infusion (Visit 7 - Week 56) | 38.74 (9.39)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.11, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.24; Mean Difference (Net) = 1.48, 95% CI 2-sided [-0.35 to 3.31] — Effect size: 0.24
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 27, analysis 1]; Test type: Other; p = 0.0046, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.24; Mean Difference (Net) = 2.69, 95% CI 2-sided [0.893 to 4.487] — Effect size: 0.24

39. Secondary Outcome: NIH Toolbox - Cognition: Pattern Comparison Processing Speed Test T Scores
Description: NIH Toolbox - Cognition: Pattern Comparison Processing Speed Test T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The NIH Toolbox consists of multiple subsections that are summed individually to create a raw score for each subsection. Then, a T-score was calculated by comparing to normative data. T-scores are standardized to have an average of 50 and a standard deviation of 10. A higher T-score indicates more of the measured construct was observed, whether it is a positive construct or a negative construct. Technically there is no minimum or maximum t-score since it is normalized.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 23
  Infusion 1/Baseline (Visit 3 - Week 0) | 30.65 (14.11)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 35.42 (17.12)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 19
  1 year Post-Infusion (Visit 7 - Week 56) | 39.68 (18.35)
Statistical Analysis 1: Comparison: HB-adMSC; Neurocognitive outcome measures will be analyzed using linear regression models to estimate differences across time points (pre- and post-treatment). Mean differences with 95% confidence intervals (CI) were determined for all outcomes at 6 and 12 months after treatment; Test type: Other; p = 0.0081, Regression, Linear — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.60; Mean Difference (Net) = 5.69, 95% CI 2-sided [1.58 to 9.77] — Effect size: 0.60
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.00017, Regression, Linear — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.60; Mean Difference (Net) = 8.505, 95% CI 2-sided [4.42 to 12.606] — Effect size: 0.60

40. Secondary Outcome: NIH Toolbox - Cognition: Picture Vocabulary Test T Scores
Description: NIH Toolbox - Cognition: Picture Vocabulary Test T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 1 year Post-Infusion (Visit 7 - Week 56). The NIH Toolbox consists of multiple subsections that are summed individually to create a raw score for each subsection. Then, a T-score was calculated by comparing to normative data. T-scores are standardized to have an average of 50 and a standard deviation of 10. A higher T-score indicates more of the measured construct was observed, whether it is a positive construct or a negative construct. Technically there is no minimum or maximum t-score since it is normalized.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 1 year Post-Infusion (Visit 7 - Week 56)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 23
  Infusion 1/Baseline (Visit 3 - Week 0) | 41.96 (8.48)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 19
  1 year Post-Infusion (Visit 7 - Week 56) | 43.74 (9.56)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.64, Regression, Linear — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.10; Mean Difference (Net) = 0.846, 95% CI 2-sided [-2.767 to 4.515] — Effect size: 0.10

41. Secondary Outcome: NIH Toolbox - Cognition: Dimensional Change Card Sort Test T Scores
Description: NIH Toolbox - Cognition: Dimensional Change Card Sort Test T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The NIH Toolbox consists of multiple subsections that are summed individually to create a raw score for each subsection. Then, a T-score was calculated by comparing to normative data. T-scores are standardized to have an average of 50 and a standard deviation of 10. A higher T-score indicates more of the measured construct was observed, whether it is a positive construct or a negative construct. Technically there is no minimum or maximum t-score since it is normalized.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 23
  Infusion 1/Baseline (Visit 3 - Week 0) | 36.65 (8.95)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 38.05 (8.57)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 19
  1 year Post-Infusion (Visit 7 - Week 56) | 40.47 (11.89)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.21, Regression, Linear — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.48; Mean Difference (Net) = 2.59, 95% CI 2-sided [-1.52 to 6.65] — Effect size: 0.48
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.040, Regression, Linear — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.48; Mean Difference (Net) = 4.318, 95% CI 2-sided [0.241 to 8.399] — Effect size: 0.48

42. Secondary Outcome: NIH Toolbox - Cognition: Franker Inhibitory Control and Attention Test T Scores
Description: NIH Toolbox - Cognition: Franker Inhibitory Control and Attention Test T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The NIH Toolbox consists of multiple subsections that are summed individually to create a raw score for each subsection. Then, a T-score was calculated by comparing to normative data. T-scores are standardized to have an average of 50 and a standard deviation of 10. A higher T-score indicates more of the measured construct was observed, whether it is a positive construct or a negative construct. Technically there is no minimum or maximum t-score since it is normalized.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 22
  Infusion 1/Baseline (Visit 3 - Week 0) | 31.68 (10.83)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 28.58 (9.81)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 19
  1 year Post-Infusion (Visit 7 - Week 56) | 31.58 (10.04)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.30, Regression, Linear — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.07; Mean Difference (Net) = -0.86, 95% CI 2-sided [-2.52 to 0.78] — Effect size: 0.07
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.33, Regression, Linear — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.07; Mean Difference (Net) = 0.789, 95% CI 2-sided [-0.83 to 2.409] — Effect size: 0.07

43. Secondary Outcome: NIH Toolbox - Cognition: List Sorting Working Memory Test T Scores
Description: NIH Toolbox - Cognition: List Sorting Working Memory Test T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The NIH Toolbox consists of multiple subsections that are summed individually to create a raw score for each subsection. Then, a T-score was calculated by comparing to normative data. T-scores are standardized to have an average of 50 and a standard deviation of 10. A higher T-score indicates more of the measured construct was observed, whether it is a positive construct or a negative construct. Technically there is no minimum or maximum t-score since it is normalized.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 23
  Infusion 1/Baseline (Visit 3 - Week 0) | 40.43 (9.61)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 39.37 (9.33)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 19
  1 year Post-Infusion (Visit 7 - Week 56) | 43.00 (10.96)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.96, Regression, Linear — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.31; Mean Difference (Net) = 0.1, 95% CI 2-sided [-3.49 to 3.66] — Effect size: 0.31
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.10, Regression, Linear — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.31; Mean Difference (Net) = 2.985, 95% CI 2-sided [-0.588 to 6.562] — Effect size: 0.31

44. Secondary Outcome: NIH Toolbox - Motor: 9-hole Pegboard Dexterity Test T Scores
Description: NIH Toolbox - Motor: 9-hole Pegboard Dexterity Test T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The NIH Toolbox consists of multiple subsections that are summed individually to create a raw score for each subsection. Then, a T-score was calculated by comparing to normative data. T-scores are standardized to have an average of 50 and a standard deviation of 10. A higher T-score indicates more of the measured construct was observed, whether it is a positive construct or a negative construct. Technically there is no minimum or maximum t-score since it is normalized.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 21
  Infusion 1/Baseline (Visit 3 - Week 0) | 26.81 (13.21)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 18
  6 months Post-Infusion (Visit 6 - Week 28) | 27.61 (13.28)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 18
  1 year Post-Infusion (Visit 7 - Week 56) | 27.94 (15.28)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.043, Regression, Linear — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.21; Mean Difference (Net) = 3.34, 95% CI 2-sided [0.13 to 6.53] — Effect size: 0.21
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.10, Regression, Linear — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.21; Mean Difference (Net) = 2.718, 95% CI 2-sided [-0.484 to 5.917] — Effect size: 0.21

45. Secondary Outcome: NIH Toolbox - Motor: 9-hole Pegboard Dexterity Test Non-Dominant Hands T Scores
Description: NIH Toolbox - Motor: 9-hole Pegboard Dexterity Test Non-Dominant Hands T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The NIH Toolbox consists of multiple subsections that are summed individually to create a raw score for each subsection. Then, a T-score was calculated by comparing to normative data. T-scores are standardized to have an average of 50 and a standard deviation of 10. A higher T-score indicates more of the measured construct was observed, whether it is a positive construct or a negative construct. Technically there is no minimum or maximum t-score since it is normalized.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 14
  Infusion 1/Baseline (Visit 3 - Week 0) | 26.21 (18.82)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 10
  6 months Post-Infusion (Visit 6 - Week 28) | 20.20 (15.06)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 11
  1 year Post-Infusion (Visit 7 - Week 56) | 25.09 (20.43)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.24, Regression, Linear — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.20; Mean Difference (Net) = 2.39, 95% CI 2-sided [-1.73 to 6.44] — Effect size: 0.20
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.061, Regression, Linear — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.20; Mean Difference (Net) = 3.79, 95% CI 2-sided [-0.152 to 7.72] — Effect size: 0.20

46. Secondary Outcome: Rey Auditory Verbal Learning Test (RAVLT) Delay T Scores
Description: Rey Auditory Verbal Learning Test (RAVLT) Delay T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The Rey Auditory Verbal Learning Test (RAVLT) Delay Test consists of calculating the total number of words recalled on the delayed recall trial (after a 20-30 minute delay). Then, a T-score is calculated by comparing to normative data adjusted for age and education to determine performance relative to peers. T-scores are standardized to have an average of 50 and a standard deviation of 10. A higher T-score indicates more words were recalled (better outcomes). Technically there is no minimum or maximum t-score since it is normalized.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 22
  Infusion 1/Baseline (Visit 3 - Week 0) | 31.95 (16.24)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 30.57 (19.02)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 19
  1 year Post-Infusion (Visit 7 - Week 56) | 37.49 (19.20)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.49, Regression, Linear — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.43; Mean Difference (Net) = 1.22, 95% CI 2-sided [-2.28 to 4.71] — Effect size: 0.43
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.00026, Regression, Linear — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.43; Mean Difference (Net) = 7.001, 95% CI 2-sided [3.506 to 10.494] — Effect size: 0.43

47. Secondary Outcome: Rey Auditory Verbal Learning Test (RAVLT) Trials 1-5 T Scores
Description: Rey Auditory Verbal Learning Test (RAVLT) Trials 1-5 T Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The Rey Auditory Verbal Learning Test (RAVLT) Trials 1-5 Test consists of calculating the total number of words correctly recalled across the five initial learning trials (Trials 1-5). Then, a T-score is calculated by comparing to normative data adjusted for age and education to determine performance relative to peers. T-scores are standardized to have an average of 50 and a standard deviation of 10. A higher T-score indicates more words were recalled (better outcomes). Technically there is no minimum or maximum t-score since it is normalized.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
t-score
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 22
  Infusion 1/Baseline (Visit 3 - Week 0) | 28.42 (14.76)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 19
  6 months Post-Infusion (Visit 6 - Week 28) | 31.01 (16.34)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 19
  1 year Post-Infusion (Visit 7 - Week 56) | 36.74 (16.94)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.083, Regression, Linear — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.61; Mean Difference (Net) = 3.98, 95% CI 2-sided [-0.51 to 8.46] — Effect size: 0.61
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.00025, Regression, Linear — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.61; Mean Difference (Net) = 9.033, 95% CI 2-sided [4.55 to 13.52] — Effect size: 0.61

48. Secondary Outcome: Wechsler Adult Intelligence Scale - IV: Coding Scaled Scores
Description: Wechsler Adult Intelligence Scale - IV: Coding Scaled Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The subsection (such as Coding) raw scores are converted into a scaled score with a mean of 10 and a standard deviation of 3. This process is standardized using age-based conversion tables. Then, these scaled scores are combined into index scores which are compared to a normative population with a standard score (mean = 100, SD = 15) to create an index score and fall into ranges of "Average" being 90-109, "High Average" 110-119, "Low Average" 80-89, "Borderline" 70-79, and "Extremely Low" below 70. Higher scores mean better outcome.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
score on a scale
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 19
  Infusion 1/Baseline (Visit 3 - Week 0) | 6.58 (3.29)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 16
  6 months Post-Infusion (Visit 6 - Week 28) | 5.88 (3.18)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 17
  1 year Post-Infusion (Visit 7 - Week 56) | 6.71 (3.69)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.53, Regression, Linear — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.20; Mean Difference (Net) = 0.25, 95% CI 2-sided [-0.55 to 1.05] — Effect size: 0.20
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.10, Regression, Linear — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.20; Mean Difference (Net) = 1.043, 95% CI 2-sided [0.284 to 1.805] — Effect size: 0.20

49. Secondary Outcome: Wechsler Adult Intelligence Scale - IV: Symbol Search Scaled Scores
Description: Wechsler Adult Intelligence Scale - IV: Symbol Search Scaled Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The subsection (such as Coding) raw scores are converted into a scaled score with a mean of 10 and a standard deviation of 3. This process is standardized using age-based conversion tables. Then, these scaled scores are combined into index scores which are compared to a normative population with a standard score (mean = 100, SD = 15) to create an index score and fall into ranges of "Average" being 90-109, "High Average" 110-119, "Low Average" 80-89, "Borderline" 70-79, and "Extremely Low" below 70. Higher scores mean better outcome.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
score on a scale
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 21
  Infusion 1/Baseline (Visit 3 - Week 0) | 6.24 (3.73)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 18
  6 months Post-Infusion (Visit 6 - Week 28) | 6.06 (2.88)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 18
  1 year Post-Infusion (Visit 7 - Week 56) | 6.83 (3.81)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.034, Regression, Linear — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.28; Mean Difference (Net) = 0.83, 95% CI 2-sided [0.07 to 1.59] — Effect size: 0.28
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.0090, Regression, Linear — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.28; Mean Difference (Net) = 1.043, 95% CI 2-sided [0.284 to 1.805] — Effect size: 0.28

50. Secondary Outcome: Wechsler Adult Intelligence Scale - IV: Processing Speed Index/Composite Scores
Description: Wechsler Adult Intelligence Scale - IV: Processing Speed Composite Scores Means and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The subsection (such as Coding) raw scores are converted into a scaled score with a mean of 10 and a standard deviation of 3. This process is standardized using age-based conversion tables. Then, these scaled scores are combined into index scores which are compared to a normative population with a standard score (mean = 100, SD = 15) to create an index score and fall into ranges of "Average" being 90-109, "High Average" 110-119, "Low Average" 80-89, "Borderline" 70-79, and "Extremely Low" below 70. Higher scores mean better outcome.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
score on a scale
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 19
  Infusion 1/Baseline (Visit 3 - Week 0) | 82.05 (17.62)
  6 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 16
  6 months Post-Infusion (Visit 6 - Week 28) | 79.44 (15.12)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 17
  1 year Post-Infusion (Visit 7 - Week 56) | 83.24 (19.23)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.13, Regression, Linear — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.25; Mean Difference (Net) = 2.8, 95% CI 2-sided [-0.84 to 6.41] — Effect size: 0.25
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.016, Regression, Linear — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.25; Mean Difference (Net) = 4.486, 95% CI 2-sided [0.938 to 8.026] — Effect size: 0.25

51. Secondary Outcome: Controlled Oral Word Association Test (COWAT) Total Scaled Scores
Description: Controlled Oral Word Association Test (COWAT) Total Scaled Scores Mean and Standard Deviations at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0), 6 months Post-Infusion (Visit 6 - Week 28), 1 year Post-Infusion (Visit 7 - Week 56). The COWAT is scored by counting the number of correct words a person produces in one minute for each of the three given letters. The total score is the sum of the unique words generated across all three trials. Higher scores are considered a better outcome. The raw total score is then compared to normative data that is based on factors such as age and education level. The scaled score has a mean of 10 and a standard deviation of 3. A t-score of < 20 indicates severe impairment.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HB-adMSC
Number analyzed (Participants) | 24
score on a scale
  Infusion 1/Baseline (Visit 3 - Week 0): number analyzed (Participants) | 17
  Infusion 1/Baseline (Visit 3 - Week 0) | 8.88 (3.26)
  Month 66 months Post-Infusion (Visit 6 - Week 28): number analyzed (Participants) | 16
  Month 66 months Post-Infusion (Visit 6 - Week 28) | 8.69 (2.30)
  1 year Post-Infusion (Visit 7 - Week 56): number analyzed (Participants) | 17
  1 year Post-Infusion (Visit 7 - Week 56) | 10.00 (2.65)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.84, Regression, Linear — [p-value comment as in outcome 26, analysis 1]; Effect size: 0.33; Mean Difference (Net) = -0.11, 95% CI 2-sided [-1.23 to 0.97] — Effect size: 0.33
Statistical Analysis 2: Comparison: HB-adMSC; [analysis description as in outcome 39, analysis 1]; Test type: Other; p = 0.053, Regression, Linear — [p-value comment as in outcome 26, analysis 2]; Effect size: 0.33; Mean Difference (Net) = 1.083, 95% CI 2-sided [-0.028 to 2.162] — Effect size: 0.33

52. Secondary Outcome: MRI Structural Measures - Global White Matter
Description: MRI Structural Measures - Global White Matter Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 114,303 (29,555)
  6 months Post-Infusion (Visit 6 - Week 28) | 108,002 (25,752)
Statistical Analysis 1: Comparison: HB-adMSC; Volumetric MRI measures were analyzed using general linear mixed models (GLMMs) to estimate differences across time points (pre- and post-treatment). Models will include time of assessment (baseline and 6 months after treatment) and baseline age as covariates with random intercepts for participants to account for within-participant correlation. Mean differences with 95% confidence intervals were determined for outcomes at 6 months after treatment; Test type: Other; p = 0.27, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -1050.25, 95% CI 2-sided [-2958.69 to 858.19]

53. Secondary Outcome: MRI Structural Measures - Global Gray Matter
Description: MRI Structural Measures - Global Gray Matter Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 430,058 (45,653)
  6 months Post-Infusion (Visit 6 - Week 28) | 427,864 (54,441)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.61, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -365.57, 95% CI 2-sided [-1835.10 to 1103.97]

54. Secondary Outcome: MRI Structural Measures - Global Corpus Callosum Matter
Description: MRI Structural Measures - Global Corpus Callosum Matter Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 836 (274)
  6 months Post-Infusion (Visit 6 - Week 28) | 757 (258)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.19, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -13.17, 95% CI 2-sided [-33.32 to 6.98]

55. Secondary Outcome: MRI Structural Measures - Hippocampus (Bilateral)
Description: MRI Structural Measures - Hippocampus (bilateral) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 6,475 (1,071)
  6 months Post-Infusion (Visit 6 - Week 28) | 6,281 (1,082)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.0072, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -32.35, 95% CI 2-sided [-54.61 to -10.09]

56. Secondary Outcome: MRI Structural Measures - Amygdala (Bilateral)
Description: MRI Structural Measures - Amygdala (bilateral) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 1,926 (457)
  6 months Post-Infusion (Visit 6 - Week 28) | 1,794 (496)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.03, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -21.88, 95% CI 2-sided [-41.11 to -2.65]

57. Secondary Outcome: MRI Structural Measures - Thalamus (Bilateral)
Description: MRI Structural Measures - Thalamus (bilateral) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 4,952 (798)
  6 months Post-Infusion (Visit 6 - Week 28) | 4,700 (778)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.061, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -42.03, 95% CI 2-sided [-85.66 to 1.61]

58. Secondary Outcome: MRI Structural Measures - Caudate (Bilateral)
Description: MRI Structural Measures - Caudate (bilateral) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 3,760 (771)
  6 months Post-Infusion (Visit 6 - Week 28) | 3,523 (636)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.18, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -39.56, 95% CI 2-sided [-98.67 to 19.56]

59. Secondary Outcome: MRI Structural Measures - Putamen (Bilateral)
Description: MRI Structural Measures - Putamen (bilateral) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 901 (1169)
  6 months Post-Infusion (Visit 6 - Week 28) | 951 (1396)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.63, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = 8.25, 95% CI 2-sided [-26.01 to 42.51]

60. Secondary Outcome: MRI Structural Measures - Pallidum (Bilateral)
Description: MRI Structural Measures - Pallidum (bilateral) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 450 (393)
  6 months Post-Infusion (Visit 6 - Week 28) | 459 (448)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.85, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = 1.47, 95% CI 2-sided [-14.84 to 17.79]

61. Secondary Outcome: MRI Structural Measures - Insula (Bilateral)
Description: MRI Structural Measures - Insula (Bilateral) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 4,985 (1,164)
  6 months Post-Infusion (Visit 6 - Week 28) | 4,772 (967)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.24, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -35.42, 95% CI 2-sided [-95.21 to 24.36]

62. Secondary Outcome: MRI Structural Measures - Hippocampus (Left)
Description: MRI Structural Measures - Hippocampus (left) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 3,180 (453)
  6 months Post-Infusion (Visit 6 - Week 28) | 3,140 (503)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.31, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -6.58, 95% CI 2-sided [-19.50 to 6.34]

63. Secondary Outcome: MRI Structural Measures - Hippocampus (Right)
Description: MRI Structural Measures - Hippocampus (right) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 3,295 (663)
  6 months Post-Infusion (Visit 6 - Week 28) | 3,141 (646)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.018, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -25.77, 95% CI 2-sided [-46.25 to -5.29]

64. Secondary Outcome: MRI Structural Measures - Amygdala (Left)
Description: MRI Structural Measures - Amygdala (left) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 870 (195)
  6 months Post-Infusion (Visit 6 - Week 28) | 813 (243)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.067, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -9.60, 95% CI 2-sided [-19.79 to 0.59]

65. Secondary Outcome: MRI Structural Measures - Amygdala (Right)
Description: MRI Structural Measures - Amygdala (right) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 1,055 (326)
  6 months Post-Infusion (Visit 6 - Week 28) | 982 (290)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.069, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -12.28, 95% CI 2-sided [-25.45 to 0.88]

66. Secondary Outcome: MRI Structural Measures - Thalamus (Left)
Description: MRI Structural Measures - Thalamus (left) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 2,522 (439)
  6 months Post-Infusion (Visit 6 - Week 28) | 2,363 (437)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.027, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -26.47, 95% CI 2-sided [-49.12 to -3.61]

67. Secondary Outcome: MRI Structural Measures - Thalamus (Right)
Description: MRI Structural Measures - Thalamus (right) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 2,431 (388)
  6 months Post-Infusion (Visit 6 - Week 28) | 2,337 (422)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.24, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -15.66, 95% CI 2-sided [-42.09 to 10.77]

68. Secondary Outcome: MRI Structural Measures - Caudate (Left)
Description: MRI Structural Measures - Caudate (left) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 1,786 (253)
  6 months Post-Infusion (Visit 6 - Week 28) | 1,679 (220)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.079, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -17.91, 95% CI 2-sided [-37.83 to 2.01]

69. Secondary Outcome: MRI Structural Measures - Caudate (Right)
Description: MRI Structural Measures - Caudate (right) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 1,974 (578)
  6 months Post-Infusion (Visit 6 - Week 28) | 1,844 (483)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.29, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -21.65, 95% CI 2-sided [-62.91 to 19.61]

70. Secondary Outcome: MRI Structural Measures - Putamen (Left)
Description: MRI Structural Measures - Putamen (left) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 224 (135)
  6 months Post-Infusion (Visit 6 - Week 28) | 199 (106)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.24, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -4.08, 95% CI 2-sided [-11.01 to 2.84]

71. Secondary Outcome: MRI Structural Measures - Putamen (Right)
Description: MRI Structural Measures - Putamen (right) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 678 (1,174)
  6 months Post-Infusion (Visit 6 - Week 28) | 752 (1,401)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.44, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = 12.33, 95% CI 2-sided [-19.69 to 44.36]

72. Secondary Outcome: MRI Structural Measures - Pallidum (Left)
Description: MRI Structural Measures - Pallidum (left) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 179 (150)
  6 months Post-Infusion (Visit 6 - Week 28) | 159 (125)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.23, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -3.25, 95% CI 2-sided [-8.67 to 2.17]

73. Secondary Outcome: MRI Structural Measures - Pallidum (Right)
Description: MRI Structural Measures - Pallidum (right) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 272 (319)
  6 months Post-Infusion (Visit 6 - Week 28) | 300 (407)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.5, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = 4.73, 95% CI 2-sided [-9.43 to 18.88]

74. Secondary Outcome: MRI Structural Measures - Insula (Left)
Description: MRI Structural Measures - Insula (left) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 2,071 (575)
  6 months Post-Infusion (Visit 6 - Week 28) | 2,016 (422)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.66, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -9.23, 95% CI 2-sided [-51.62 to 33.16]

75. Secondary Outcome: MRI Structural Measures - Insula (Right)
Description: MRI Structural Measures - Insula (right) Volumes Mean and Standard Deviation at the following timepoints: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28). SupraMD is a type of mean diffusivity MRI that uses water diffusion within brain tissue to measure volume of various types of brain matter in mm3.
Time Frame: Infusion 1/Baseline (Visit 3 - Week 0) and 6 months Post-Infusion (Visit 6 - Week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SupraMD volume (mm3)
Arm/Group | HB-adMSC
Number analyzed (Participants) | 20
SupraMD volume (mm3)
  Infusion 1/Baseline (Visit 3 - Week 0) | 2,914 (748)
  6 months Post-Infusion (Visit 6 - Week 28) | 2,756 (688)
Statistical Analysis 1: Comparison: HB-adMSC; [analysis description as in outcome 52, analysis 1]; Test type: Other; p = 0.24, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Net) = -26.19, 95% CI 2-sided [-70.22 to 17.84]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of consent until the subject completed the final study visit or until the subject (or LAR) prematurely withdrew from participation (Week 0 to Week 108 - Screening to Follow-Up Call #2)
Arm/Group | HB-adMSC
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 24/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HB-adMSC (N=24)
COVID-19 Infection (Infections and infestations) | 4 (4)
Cold intolerance (General disorders) | 1 (1)
Decreased sensitivity, left side of face (Nervous system disorders) | 1 (1)
Depression, worsening (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Eosinophil count increased (Blood and lymphatic system disorders) | 1 (1)
Fall (Nervous system disorders) | 3 (4)
Fatigue, increased (General disorders) | 1 (1)
Gait disturbance (Nervous system disorders) | 1 (1)
Head cold (General disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hypoglycemia (Blood and lymphatic system disorders) | 2 (7)
Insomnia (Nervous system disorders) | 1 (1)
Itchiness, face, left side (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Motor vehicle collision (General disorders) | 1 (1)
Pain, back (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain, generalized joint and muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, tongue (Musculoskeletal and connective tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (5)
Spasticity, left arm, increased, intermittent (Nervous system disorders) | 1 (1)
Strabismus eye surgery (Eye disorders) | 1 (1)
Urinary Tract Infection symptoms (Renal and urinary disorders) | 1 (1)
Vision, worsening, intermittent (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT04063215/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT04063215/SAP_004.pdf
  • Informed Consent Form: English (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT04063215/ICF_002.pdf
  • Informed Consent Form: Spanish (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT04063215/ICF_003.pdf